CLINICAL TRIAL: NCT06591585
Title: Midterm Follow up of Pediatric Pelvic Fracture Management at Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kirollos Raafat Ramzy Wahba, doctor, Assiut University
Other Study IDs: MFU pediatric pelvic fracture
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fracture Healing
Keywords: pediatric pelvic fracture
MeSH Terms: interventions — Fracture Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Fracture Healing — A-Clinical evaluation
  1. Patients will be recruited for evaluation of documented short / long term complications:
     * subcutaneous haematoma
     * pin tract infection
     * surgical site infection
     * limb length discrepancy
     * arthritis of the hip and spine
     * SI joint pain or fusion
     * scoliosis
  2. Visually assisted gait analysis B- Radiographic evaluation
  1-Radiographic evaluation of pelvic integrity by plain X-ray ( Antero-posterior . inlet . outlet views) 2- Long film for limb length discrepancy 3- plain x ray whole spine Anterior -posterior & lateral for scoliosis

SUMMARY:
Midterm radiographic and function follow up of pediatric pelvic fractures managed at Assiut University Hospital ( AUH) with a minimum of 3 years Analysis of all recorded cases of pediatric Pelvic Fracture in AUH trauma unit from 2015 until june 2024

DETAILED DESCRIPTION:
Pelvic fractures in children as a result of trauma are uncommon and typically follow high-energy trauma [1].

Due to flexible sacroiliac joints (SIJs) and symphysis pubis, the young pediatric skeleton has inherent flexibility, which makes pediatric pelvic fractures (PPFs) different from adult pelvic fractures . Additionally, the cartilaginous cover serves as a shock absorber. [2].

Since the young skeleton can remodel , nonsurgical therapy has been the norm for PPF; nevertheless, this has resulted in a number of long-term problems, such as nonunion, malunion, scoliosis, and pelvic asymmetry. Children with unstable pelvic fractures may experience chronic neurological impairment, low back pain, persistent pain, and limping in up to 30% of cases [2]. Several factors determine whether to treat these fractures surgically or nonsurgically: Initially, the physiological age of the patient AO/OTA classification, divides pelvic fractures into three basic types

. Type A pelvic fractures does not involve the posterior arch (stable), whereas type B results from rotational forces that cause partial posterior complex disruption (rotationally unstable). In type C, there is complete posterior complex disruption (rotationally and vertically unstable).

According to a study established by the German Trauma Society (DGU) and the German Section of the Association for Osteosynthesis /Association for the Study of Internal Fixation (AO/ASIF) International in 1991. The registry provides data on all patients suffering pelvic fractures within a 14-year time frame. They identified a total of 9684 patients including 1433 pelvic fractures in children aged ≤17 years , in pelvic factures of Type A (Tile classification of pelvic fractures), a standard mortality ratio (SMR)( The standardized mortality ratio is the ratio of observed deaths in the study group to expected deaths in the general population) of 0.76 was recorded, in Type B fractures 0.65, and in Type C fractures 0.79. [3].

In our institute, Assiut University Hospital Trauma Unit, pelvic fracture cases were recorded from 2015 until june 2023 , 2041 cases of pelvic fracture were recorded 222 of those cases belong to age group below 17 years so pediatric pelvic fractures represent 10.87% of all recorded pelvic fractures.

The main question in our research proposal according to protocol discussion is what happens after pelvic fracture in pediatric cases as regards to deformities and can remodelling in pediatrics fix these deformities and what is the effect of these deformities on function later on

ELIGIBILITY:
Inclusion Criteria:

1. patient age ≤17years
2. Open fracture\ Closed fractures
3. with or without neurovascular injury
4. polytrauma (including femur & tibia fracture)
5. patients who were treated conservatively (bed rest + traction)
6. patients treated surgically

Exclusion Criteria:

* patients aged >17 years Isolated acetabulum Fractures Sample size calculation : Sample size was calculated using Epi- Info7. According to results of previous study [4] , Pelvic asymmetry occurs in 9.2% of patients undergoing open reduction internal fixation . Based on this percentage, confidence limits of 5% and a confidence level of 95%, the sample needed for the study was estimated to be about 63 patients

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with age ≤17years with Open fracture\ Closed fractures pelvis that was treated surgically or not
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Modified Majeed Functional scoring system | base line

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sanz-Esteban I, Calvo-Lobo C, Rios-Lago M, Alvarez-Linera J, Munoz-Garcia D, Rodriguez-Sanz D. Mapping the human brain during a specific Vojta's tactile input: the ipsilateral putamen's role. Medicine (Baltimore). 2018 Mar;97(13):e0253. doi: 10.1097/MD.0000000000010253. PMID 29595683